CLINICAL TRIAL: NCT06187987
Title: Outcomes of Mechanical Thrombectomy With the FlowTriever Device in Acute Pulmonary Embolism, Results of a Swedish Retrospective Analysis
Brief Title: Mechanical Thrombectomy With the FlowTriever Device in Acute Pulmonary Embolism - a Retrospective Analysis
Status: Completed | Type: Observational
Sponsor: Kristina Svennerholm (Other)
Collaborators: Stockholm South General Hospital (Other); Karolinska University Hospital (Other); Danderyd Hospital (Other); University Hospital, Linkoeping (Other); Sunderby Hospital (Other)
Responsible Party: Sponsor-Investigator, Kristina Svennerholm, Principal investigator. MD. PhD., Sahlgrenska University Hospital
Organization: Sahlgrenska University Hospital (Other)
Other Study IDs: Flow-PE
Record Dates: First submitted 2023-12-12; First posted 2024-01-03 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Pulmonary Embolism
Keywords: FlowTriever; Catheter-Directed Intervention; Aspirational thrombectomy
MeSH Terms: conditions — Pulmonary Embolism | interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- FlowTriever: Acute PE patients treated with the FlowTriever device
  Interventions: Device: Mechanical thrombectomy
- Intravenous Thrombolysis: Acute PE patients treated with intravenous thrombolysis
  Interventions: Drug: Intravenous thrombolysis

INTERVENTIONS:
Device: Mechanical thrombectomy — Aspirational mechanical thrombectomy
  Other Names: FlowTriever
  Groups: FlowTriever
Drug: Intravenous thrombolysis — Intravenous thrombolysis with tissue-type plasminogen activator (tPA)
  Other Names: Alteplase
  Groups: Intravenous Thrombolysis

SUMMARY:
International guidelines recommend intravenous thrombolysis (IVT) for high-risk pulmonary embolism (PE). In high-risk PE where IVT is contraindicated or has failed, surgical embolectomy or catheter-directed intervention (CDI) is recommended. CDI is also recommended as an alternative in patients with intermediate-risk PE with haemodynamic deterioration during anticoagulation treatment.

Although there is a lack of randomized studies comparing CDI to anticoagulation or systemic thrombolysis in PE, several studies and recent meta-analyses have shown that CDI is an effective treatment that is associated with fewer complications than IVT, especially bleeding.

DETAILED DESCRIPTION:
The FlowTriever® retrieval/aspiration system is the first mechanical thrombectomy device to receive PE as an indication from the United States Food and Drug administration agency. It combines large-bore aspiration with expanding mesh disks designed to trap and subsequently retract the blood clots from the pulmonary arteries. While Inari Medical, the medical device company that produces the FlowTriever® system, has initiated and published a few prospective trials on FlowTriever® in PE, non-industry sponsored studies are small and mostly retrospective.

In 2021 FlowTriever® became the primary device for CDI in PE at Sahlgrenska University Hospital in Gothenburg, Sweden. Concurrently, several hospitals in Sweden have started using FlowTriever® in high-risk PE. As such, the method needs evaluation and validation on a local and national level.

This retrospective observational study aims to evaluate the outcomes of patients with acute PE treated with the FlowTriever® device in Sweden. A control group consisting of PE patients treated with IVT will be used for comparison.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Acute PE verified by computed tomography (CT) or angiography
* PE treated with thrombolysis or FlowTriever® during the time period from January 1st of the year when FlowTriever was introduced at each respective participating center to the end of 2023.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with acute PE
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Composite endpoint of survival and major bleeding | up to 7 days and up to 30 days
  Composite endpoint of survival at 30 days and major bleeding within 7 days, after intervention.

SECONDARY OUTCOMES:
Survival | up to 30 days
  Survival at 30 days.
Major Bleeding | up to 7 days
  Major bleeding within 7 days after intervention.
Right Ventricle/Left Ventricle (RV/LV) ratio | from 48 hours before intervention up to 48 hours after intervention
  Change in RV/LV-ratio with the intervention.
Total Length of stay in the ICU or IMCU | From administration until discharge from ICU/IMCU, up to 30 days
  Length of stay in the ICU/IMCU
Total Length of stay in hospital | From diagnosis of PE until discharge from hospital, up to 30 days
  Length of stay in hospital

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Svennerholm, MD, PhD, Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-03-16): https://cdn.clinicaltrials.gov/large-docs/87/NCT06187987/SAP_000.pdf